CLINICAL TRIAL: NCT06943911
Title: Empowering Breast Cancer Clients Through AI Chatbots: Transforming Knowledge and Attitudes for Enhanced Nursing Care
Brief Title: Reflects the Intervention (AI Chatbot)
Acronym: BC-CHAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mostafa Shaban (Other)
Responsible Party: Sponsor-Investigator, Mostafa Shaban, Dr, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KFSU-BC-AI-2025
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: AI Chatbot; Breast Cancer; Patient Education; Empowerment; Oncology Nursing; Attitudes Toward AI; Digital Health; Patient Support
MeSH Terms: conditions — Breast Neoplasms; Empowerment

STUDY DESIGN:
Intervention Model Description: This study uses a quasi-experimental, parallel group design, where one group receives an AI chatbot intervention alongside standard care, while the other group receives only standard care. The groups will be compared to measure the intervention's effectiveness on knowledge improvement, AI attitudes, and empowerment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (AI Chatbot + Standard Care) (Experimental): Participants in this arm will receive standard oncology care in addition to interacting with an AI-powered chatbot. The chatbot will provide personalized educational content on breast cancer, treatment options, side effects, and offer emotional support. Participants will engage with the chatbot for 4 weeks, with assessments at baseline and post-interventi
  Interventions: Behavioral: AI Chatbot for Breast Cancer Patient Education and Empowerment
- Control Group (Standard Care Only) (No Intervention): Participants in this arm will receive standard oncology care only, including routine consultations with oncology specialists and nurses. They will not have access to the AI chatbot intervention.

INTERVENTIONS:
Behavioral: AI Chatbot for Breast Cancer Patient Education and Empowerment — The AI Chatbot for Breast Cancer Patient Education and Empowerment is a digital health intervention that leverages artificial intelligence to provide personalized educational content and emotional support to breast cancer patients. The chatbot delivers information on breast cancer management, treatment options, side effects, and self-care practices. It is available 24/7, offering real-time answers to patient queries and tailored suggestions based on their treatment path. The aim is to increase patient knowledge, improve attitudes toward AI, and empower patients to take a more active role in their care. The chatbot intervention is provided alongside standard oncology care at Kafr El-Sheikh University Hospital.
  Arms: Intervention Group (AI Chatbot + Standard Care)

SUMMARY:
The goal of this clinical trial is to investigate the impact of an AI-powered chatbot intervention on improving knowledge, attitudes, and empowerment in breast cancer patients. The study focuses on female breast cancer patients, aged 18 years or older, who are receiving treatment at Kafr El-Sheikh University Hospital in Egypt.

The main questions it aims to answer are:

Can the AI chatbot intervention improve breast cancer knowledge compared to standard care?

Can the AI chatbot intervention positively influence attitudes toward AI in healthcare?

Does the AI chatbot intervention enhance patient empowerment in managing breast cancer?

Researchers will compare:

Intervention group (AI chatbot + standard care) to control group (standard care alone) to see if the AI chatbot intervention leads to greater improvements in knowledge, more positive attitudes towards AI, and higher perceived empowerment.

Participants will:

Engage with an AI-powered chatbot designed to provide personalized education on breast cancer, treatment options, and emotional support.

Complete pre- and post-intervention assessments to measure changes in knowledge, attitudes toward AI, and empowerment.

Receive standard care, including routine oncology consultations and nursing support, alongside the chatbot intervention (for the intervention group).

DETAILED DESCRIPTION:
This study explores the integration of AI-powered chatbots in breast cancer care to enhance patient education, self-management, and psychosocial support. Breast cancer is often accompanied by a range of psychological challenges, including anxiety and uncertainty about treatment options, side effects, and overall prognosis. Traditional healthcare systems struggle to provide continuous support, which is where AI technology can offer a solution by enabling 24/7 access to information and emotional support.

The study design employs a quasi-experimental approach, where 122 breast cancer patients were recruited from Kafr El-Sheikh University Hospital. Participants were randomly assigned to one of two groups:

Intervention Group (n=61): Participants in this group received standard care, which includes routine consultations with oncology specialists and nurses, in addition to an AI chatbot intervention. The chatbot delivered personalized educational content about breast cancer, treatment options, and self-care. It also offered emotional support by answering queries and providing motivational messages.

Control Group (n=61): Participants in this group received only standard care, which consisted of regular oncology consultations and nursing support without the chatbot.

The AI chatbot intervention is designed to:

Improve knowledge about breast cancer, treatment side effects, symptom management, and emotional well-being.

Foster positive attitudes toward AI in healthcare by providing a reliable, non-judgmental source of information.

Enhance empowerment by allowing patients to actively engage with their care information outside of regular hospital visits.

Participants' knowledge, attitudes toward AI, and empowerment were assessed at two time points:

Baseline (before the intervention)

Post-intervention (after 4 weeks of engaging with the chatbot)

The primary outcome of the study is to evaluate improvements in breast cancer-related knowledge, measured through a questionnaire that assesses knowledge in key areas such as early detection, treatment options, side effects, and AI's role in healthcare. The secondary outcomes focus on attitudes toward AI and perceived empowerment, assessed through validated Likert scales designed for this purpose.

This study will provide valuable insights into the feasibility and efficacy of AI-powered chatbots in enhancing patient care for breast cancer patients, especially in resource-limited settings. Furthermore, it aims to contribute to the growing body of evidence supporting the use of digital health technologies in oncology nursing and patient empowerment.

ELIGIBILITY:
Inclusion Criteria:

Female participants diagnosed with breast cancer, regardless of cancer stage.

Age 18 years or older.

Ability to read and communicate in Arabic to interact with the AI chatbot.

Willingness to participate in the study and to engage with the AI chatbot for the duration of the intervention.

Ability to provide informed consent.

Exclusion Criteria:

Participants with cognitive impairments or serious mental health conditions that may hinder understanding or participation in the study.

Patients currently receiving palliative care, as they may prioritize symptom management over educational interventions.

Participants who are physically unable to engage with the study's digital tools or complete assessments (e.g., due to severe illness).

Individuals who are unable to communicate in Arabic, as the AI chatbot intervention is designed in Arabic.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Breast Cancer Knowledge Improvement | 2 months
  This outcome measures the change in breast cancer knowledge from baseline to post-intervention for participants who used the AI chatbot compared to the control group. Knowledge is assessed using the Artificial Intelligence of Breast Cancer Questionnaire, which covers topics such as treatment options, side effects, symptom management, and AI's role in healthcare.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
We currently do not plan to share individual participant data (IPD) outside of the research team due to concerns about participant confidentiality and the sensitive nature of the data collected. The study includes personal health information that is protected under ethical guidelines and privacy regulations. Additionally, sharing IPD may present challenges related to data security and informed consent, as participants have not explicitly consented to broader data sharing. However, the study's aggregate findings will be made publicly available through peer-reviewed publications and presentations

REFERENCES:
- [Background] Janopaul-Naylor JR, Koo A, Qian DC, McCall NS, Liu Y, Patel SA. Physician Assessment of ChatGPT and Bing Answers to American Cancer Society's Questions to Ask About Your Cancer. Am J Clin Oncol. 2024 Jan 1;47(1):17-21. doi: 10.1097/COC.0000000000001050. Epub 2023 Oct 12. PMID 37823708
- [Background] Siglen E, Vetti HH, Lunde ABF, Hatlebrekke TA, Stromsvik N, Hamang A, Hovland ST, Rettberg JW, Steen VM, Bjorvatn C. Ask Rosa - The making of a digital genetic conversation tool, a chatbot, about hereditary breast and ovarian cancer. Patient Educ Couns. 2022 Jun;105(6):1488-1494. doi: 10.1016/j.pec.2021.09.027. Epub 2021 Oct 6. PMID 34649750
- [Background] Agrawal A. Fairness in AI-Driven Oncology: Investigating Racial and Gender Biases in Large Language Models. Cureus. 2024 Sep 16;16(9):e69541. doi: 10.7759/cureus.69541. eCollection 2024 Sep. PMID 39416584
- [Background] Ma Y, Achiche S, Pomey MP, Paquette J, Adjtoutah N, Vicente S, Engler K; MARVIN chatbots Patient Expert Committee; Laymouna M, Lessard D, Lemire B, Asselah J, Therrien R, Osmanlliu E, Zawati MH, Joly Y, Lebouche B. Adapting and Evaluating an AI-Based Chatbot Through Patient and Stakeholder Engagement to Provide Information for Different Health Conditions: Master Protocol for an Adaptive Platform Trial (the MARVIN Chatbots Study). JMIR Res Protoc. 2024 Feb 13;13:e54668. doi: 10.2196/54668. PMID 38349734
- [Background] Chang YC, Wu CH, Lupo R, Botti S, Conte L, Vitone M, Massafra R, De Nunzio G, Vitale E. Generative Artificial Intelligence (AI) to Uncover Insights From Breast Cancer Patients' Perceptions to Mindfulness-Based Stress Reduction (MBSR) Interventions. Holist Nurs Pract. 2025 Sep-Oct 01;39(5):317-325. doi: 10.1097/HNP.0000000000000677. Epub 2025 Aug 13. PMID 39186509
- [Background] Sato A, Haneda E, Hiroshima Y, Narimatsu H. Preliminary Screening for Hereditary Breast and Ovarian Cancer Using an AI Chatbot as a Genetic Counselor: Clinical Study. J Med Internet Res. 2024 Nov 27;26:e48914. doi: 10.2196/48914. PMID 39602801
- [Derived] Shaban M, Osman YM, Mohamed NA, Shaban MM. Empowering breast cancer clients through AI chatbots: transforming knowledge and attitudes for enhanced nursing care. BMC Nurs. 2025 Jul 29;24(1):994. doi: 10.1186/s12912-025-03585-w. PMID 40731340